CLINICAL TRIAL: NCT02179645
Title: A Three-Part, Phase I Study Of Orally Administered GRC 27864, A Novel, Microsomal Prostaglandin E Synthase-1 Enzyme (mPGES-1) Inhibitor, To Evaluate The Safety, Tolerability And PK Of Single Ascending Doses In Healthy, Adult Subjects (Part 1a), And Of A Single Dose In Elderly Subjects (Part 2); The Effect Of Food On PK (Part 1b) In Healthy, Adult Subjects; And To Compare The Effects On Prostanoid Metabolism With Celecoxib (Part 3) In Healthy, Adult Subjects.
Brief Title: GRC 27864 First in Man, Single Ascending Dose Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Glenmark Pharmaceuticals Ltd. India (Industry)
Collaborators: Glenmark Pharmaceuticals S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: GRC 27864-101
Record Dates: First submitted 2014-06-26; First posted 2014-07-02 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- GRC 27864 (Experimental): Test Treatment GRC 27864
  Interventions: Drug: GRC 27864
- Celecoxib (Active Comparator): Active Comparator Treatment
  Interventions: Drug: Celecoxib
- Placebo (Placebo Comparator): Placebo Treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GRC 27864
  Arms: GRC 27864
Drug: Celecoxib
  Arms: Celecoxib
Drug: Placebo
  Arms: Placebo

SUMMARY:
A Single Dose Study of GRC 27864 in Healthy Volunteers.

DETAILED DESCRIPTION:
This is a phase I study of GRC 27864 in healthy volunteers. The purposes of this study are to look at safety, how well the study drug is tolerated, how much of the study drug gets into the blood stream, and how long it takes the body to get rid of it when given to humans. Information about any side effects that may occur will also be collected. Participants will remain in the study for approximately 3 months. This study is for research purposes only and is not intended to treat any medical condition.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female healthy subjects, age ≥18 to ≤55 years (≥65 years for elderly subjects study) at the time of informed consent
2. Body mass index between 18.5 and 32.0 kilograms per square meter (kg/m2), inclusive
3. Female subjects who are of child-bearing potential or had tubal ligation must agree to use highly effective methods of contraception
4. Male subjects whose partners are of child-bearing potential or had tubal ligation must also agree to use two highly effective method of contraception

Exclusion Criteria:

1. Subjects with inherited or acquired disorders in platelet function, bleeding or coagulation.
2. Presence of any clinically relevant acute or chronic disease which could interfere with the subject safety during the clinical study, expose the subject to undue risk.
3. Veins unsuitable for repeat venepuncture.
4. Presence of clinical laboratory test values judged clinically significant by the investigator.
5. Positive test results for hepatitis B surface antigen (HBsAg), hepatitis C virus antibodies (HCVAb) or human immunodeficiency virus (HIV)-1 and/or -2 antibodies at screening.
6. History or presence of drug abuse at screening or upon admission to the CRU.
7. Participation in another clinical study with an experimental drug within 3 months before the first administration of the IMP.
8. Any psychological, emotional problems, any disorders or resultant therapy that is likely to invalidate informed consent, or limit the ability of the subject to comply with the Clinical Study Protocol requirements.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2014-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Drug related adverse events (AEs) or any serious AEs | 15 days after administration of the study drug
  All treatment-emergent adverse events (TEAE) occurring in the study, in terms of nature, onset, duration, severity, relationship and outcome of adverse events and serious adverse events, in adult healthy volunteers from baseline to day 15.

SECONDARY OUTCOMES:
Time to Maximum Concentration (Tmax) of GRC 27864 | Pre-dose to and post-dose from 15 minutes to 72 hours
Maximum Concentration (Cmax) of GRC 27864 | Post dose up to 72 hours
Area Under Curve [(AUC (0-∞) and AUC (0-t)] of GRC 27864 | Pre-dose to and post-dose from 15 minutes to 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jim Bush, MB ChB, Principal Investigator — Medical Director
Locations (1):
- Covance Clinical Research Unit, Leeds, Yorkshire, United Kingdom